CLINICAL TRIAL: NCT07211516
Title: Improving Workforce Participation and Well-Being in Individuals With Multiple Sclerosis
Brief Title: Relationship Between Cognition, Workforce Participation and Well-Being in Individuals With Multiple Sclerosis
Status: Not yet recruiting | Type: Observational
Sponsor: Region Gävleborg (Other)
Collaborators: University of Gavle (Other)
Responsible Party: Sponsor
Other Study IDs: MSCogWork2
Record Dates: First submitted 2025-09-22; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-09

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with MS and of working age (18-65) who have been referred to neuropsychological evaluation.: Time of neuropsychological assessment from 5 years before until study start.

SUMMARY:
Multiple sclerosis (MS) is a chronic neurodegenerative disease and a leading cause of reduced workforce participation due to neurological illness in Western countries. Over the past 30 years, new treatments have reduced symptom burden, allowing patients to stay in the workforce longer. However, fatigue and cognitive impairments remain major barriers to work capacity. This project aims to examine factors important for work ability and well-being in persons with MS and cognitive impairments. The specific research questions are:

1. How do job type and opportunities for workplace adaptations influence work ability and well-being in individuals with MS and cognitive impairments?
2. What are the associations between cognitive function in MS and work ability as well as well-being? The investigators plan to collect data on patients with MS who have undergone a neuropsychological assessment at the neurology clinic in Region Gävleborg over a five year period. Approximately 100 patients are eligible for participation. Data will be collected through surveys and by extracting information from medical records. The surveys include questions related to well-being and work ability. Data from medical records contain data from the neuropsychological assessment, other rehabilitation interventions as well as data related to treatment and progress of MS.

The findings from the study aim to enhance work-oriented rehabilitation and provide a deeper understanding of how to support individuals with MS in maintaining employment and overall well-being

ELIGIBILITY:
Inclusion Criteria:

Multiple sclerosis Age between 18-65 Performed a neuropsychological assessment at the Neurology department at Gävle Hospital during the last 5 years (counting from study start) -

Exclusion Criteria:

Other diagnosis hindering work participation more than MS

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of working age with MS in Region Gävleborg who have performed a neuropsychological assessment during the 5 years prior to study start and who are not suffering from other diagnosis which impact their work ability to a large extent.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Work participation | Baseline
  Percentage of full-time work. 100 % full-time work and 0% is not working at all.
Hospital anxiety and depression scale (HADS) | Baseline
  Self-assessment of anxiety and depression. Consists of two scales measuring the probability of having anxiety and depression respectively. Min score 0, max 21 for each scale. Higher scores indicate higher probability of anxiety/depression.
WHO-5 Well-Being Index | Baseline
  Overall rating of well-being. The WHO-5 score range is a raw score of 0-25, which is then multiplied by 4 to get a percentage score of 0-100. Higher score indicates higher well-being.
Brief index of job satisfaction (BIAJS) | Baseline
  The Brief Index of Affective Job Satisfaction (BIAJS) has a score range of 1 to 5 for each of its four items, based on a 5-point Likert scale where 1 is "strongly disagree" and 5 is "strongly agree". The total BIAJS score is the sum of these four items, resulting in a possible range from 4 to 20, with higher scores indicating greater affective job satisfaction.

SECONDARY OUTCOMES:
Work-life balance | Baseline
  Questions from the subscale "Quantitative demands" of the Copenhagen Psychosocial Questionnaire (COPSOQ-III) related to the demands of work. The COPSOQ-III uses Likert-like scales, and its items are coded with values of 0, 25, 50, 75, and 100 to achieve a 0-100 scale. Higher scores indicate more demands.
Can-Work-S | Baseline
  Three questions from a questionnaire developed to measure work-life balance after cancer. Each item ranges from 1 to 5 with higher scores indicating worse work-life balance.

CONTACTS AND LOCATIONS:
Locations (1):
- Gävle hospital, Gävle, Sweden

IPD SHARING:
Plan to Share IPD: No
To comply with the conditions set by the ethical review board, individual participant data (IPD) cannot be shared with other researchers. However, aggregated data are available upon reasonable reques